CLINICAL TRIAL: NCT02461771
Title: Assessment of Safety, Tolerability and Pharmacokinetics of Intravitreal APL-2 Therapy for Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Assessment of Safety, Tolerability and Pharmacokinetics of Intravitreal Pegcetacoplan (APL-2) for Patients With Wet AMD
Acronym: ASAP II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: POT-CP043014
Record Dates: First submitted 2015-06-02; First posted 2015-06-03 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: AMD; Wet AMD; Neovascular AMD
MeSH Terms: interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pegcetacoplan Cohort 1 (Experimental): 4 mg of pegcetacoplan 100 μL IVT injection
  Interventions: Drug: Pegcetacoplan
- Pegcetacoplan Cohort 2 (Experimental): 10 mg of pegcetacoplan 100 μL IVT injection
  Interventions: Drug: Pegcetacoplan
- Pegcetacoplan Cohort 3 (Experimental): 20 mg of pegcetacoplan 100 μL IVT injection
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — On treatment day, subjects will be administered a single 100 μL IVT injection of pegcetacoplan at the dose corresponding to their treatment assignment.
  Other Names: APL-2

SUMMARY:
The objective of this study is to provide initial safety, tolerability and pharmacokinetics information of intravitreal administration of pegcetacoplan in order to support further development into larger Phase II studies for treatment of patients with AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age ≥ 50 years
3. The presence of an active choroidal neovascular lesion secondary to AMD
4. On treatment with anti-VEGF therapy (Lucentis®, Eylea® or Avastin®)
5. Must have received at least 3 anti-VEGF treatments over the 26-week period prior to screening (Screening Visit)
6. Evidence that the macular fluid has responded to anti-VEGF in the past based on OCT in the opinion of PI
7. At screening, evidence of subretinal fluid and retinal cystic changes
8. Must have received anti-VEGF treatment within 10 days prior to pegcetacoplan treatment (anti-VEGF can be administered on the same day of the screening visit after the screening procedures have been completed)
9. OCTs of sufficient quality to allow for the assessment of the central macular fluid can be obtained
10. Female subjects must be:

    * Women of non-child-bearing potential (WONCBP), Or
    * Women of child-bearing potential (WOCBP) with a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study
11. Males with female partners of child-bearing potential must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study
12. Willing and able to give informed consent

Exclusion Criteria:

1. Choroidal neovascularization associated with other ocular diseases such as pathologic myopia, ocular histoplasmosis or posterior uveitis, etc
2. Decreased vision due to retinal disease not attributable to choroidal neovascularization, such as nonexudative forms of AMD, geographic atrophy, inherited retinal dystrophy, uveitis or epiretinal membrane, a vitelliform-like lesion of the outer retina (e.g., as in pattern dystrophies or basal laminar drusen), idiopathic parafoveal telangiectasis, or central serous retinopathy
3. Additional ocular diseases that have irreversibly compromised or, during follow-up, could likely compromise the VA of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non proliferative diabetic retinopathy, or proliferative diabetic retinopathy
4. Decreased vision due to significant media opacity such as corneal disease or cataract, or opacity precluding photography of the retina
5. Cataract surgery within three months of enrollment
6. Presence of any hemorrhage
7. History of treatment for CNV:

   1. Previous PDT treatment within 30 days prior to enrollment in the study
   2. Previous extrafoveal or juxtafoveal thermal laser photocoagulation within 30 days prior to enrollment in the study
8. Intraocular surgery (including lens replacement surgery) within 3 months prior to randomization
9. Medical problems that make consistent follow-up over the treatment period unlikely (e.g. stroke, severe MI, end stage malignancy), or in general a poor medical risk because of other systemic diseases or active uncontrolled infections
10. Hypersensitivity to fluorescein

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2016-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Grossi, MD PhD, Study Director — Apellis Pharmaceuticals, Inc.
Locations (4):
- United States (3):
  - United States, California, Beverly Hills, California
  - United States, Florida, Miami, Florida
  - United States, New Hampshire, Portsmouth, New Hampshire
- Australia, New South Wells, Parramatta, New South Wales, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female subjects aged at least 50 years with the presence of an active choroidal neovascular lesion secondary to age-related macular degeneration were recruited to this Phase 1 open-label, single-dose escalation study at 4 study centers in the United States and Australia.
Pre-assignment Details: Subjects had received at least 3 anti-vascular endothelial growth factor treatments over the 26 week period prior to screening, and were enrolled into 1 of 3 cohorts to receive pegcetacoplan (previously known as APL-2). If both eyes were eligible for the study, the subject and Principal Investigator chose the eye that served as the study eye.
Groups:
- Cohort 1: 4 milligrams (mg) pegcetacoplan: Subjects received a single intravitreal (IVT) injection of pegcetacoplan (100 microliters [μL] of 40 mg per milliliter [mg/mL]) on Day 1.
- Cohort 2: 10 mg pegcetacoplan: Subjects received a single IVT injection of pegcetacoplan (100 μL of 100 mg/mL) on Day 1.
- Cohort 3: 20 mg pegcetacoplan: Subjects received a single IVT injection of pegcetacoplan (100 μL of 200 mg/mL) on Day 1.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 3 | 3 | 7
Completed (Completed acute safety observation period (up to Day 15) and follow-up visits up to Day 113.) | 3 | 3 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all subjects who received any amount of study drug.
Groups:
- Cohort 1: 4 mg pegcetacoplan: Subjects received a single IVT injection of pegcetacoplan (100 μL of 40 mg/mL) on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 3 | 7 | 13
Age, Continuous [Median (Full Range); unit: years] | 70 [60 to 73] | 79 [74 to 81] | 72 [68 to 93] | 73 [60 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 8
  Male | 2 | 1 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 7 | 13
  Hispanic or Latino | 0 | 1 | 2 | 3
  Non-Hispanic or Latino | 3 | 2 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Ocular and Systemic Adverse Events (AEs), Including by Severity
Description: Safety was assessed throughout the study. A TEAE was defined as any AE that started on/after the IVT injection of pegcetacoplan.
Time Frame: Day 1 to Day 113
Population: The safety set included all subjects who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
Participants
  All TEAEs | 2 | 2 | 4
  Ocular TEAEs | 1 | 1 | 2
  Treatment-related AEs | 0 | 0 | 2
  Serious AEs | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0

2. Primary Outcome: Number of Dose Limiting Toxicities (DLTs)
Description: The occurrence of any of the following AEs were considered DLTs: intraocular inflammation (vitritis or uveitis), endophthalmitis, sustained elevation of intraocular pressure ≥30 millimeters (mm) of mercury, and/or sustained loss of visual acuity ≥15 letters not attributable to the injection procedure or progression of disease.
Time Frame: Day 1 to Day 15
Population: The safety set included all subjects who received any amount of study drug.
Measure: Number; unit: Number of DLTs
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
Number of DLTs | 0 | 0 | 0

3. Primary Outcome: Median Area Under the Serum Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC[0-t])
Description: The AUC(0-t) was measured using the linear trapezoidal method when concentrations were increasing and the logarithmic trapezoidal method when concentrations were decreasing. The median AUC(0-t) is presented for each cohort.
Time Frame: Predose (screening), postdose Day 3 to Day 113
Population: The pharmacokinetic (PK) set included all subjects in the safety set who had at least one postdose PK sample drawn with a measurable serum concentration of the study drug (even if the concentration was < lower limit of quantification).
Measure: Median (Full Range); unit: micrograms*day/milliliter (μg*day/mL)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
micrograms*day/milliliter (μg*day/mL) | 11.89 [11.49 to 13.90] | 29.95 [24.27 to 53.59] | 69.53 [55.06 to 86.92]

4. Primary Outcome: Median Dose Normalized AUC(0-t)
Description: The AUC(0-t) was measured using the linear trapezoidal method when concentrations were increasing and the logarithmic trapezoidal method when concentrations were decreasing. The dose normalized AUC(0-t) was calculated for each subject by dividing the parameter by the subject's respective dose in milligrams. The median dose normalized AUC(0-t) is presented for each cohort.
Time Frame: Predose (screening), postdose Day 3 to Day 113
Population: The PK set included all subjects in the safety set who had at least one postdose PK sample drawn with a measurable serum concentration of the study drug (even if the concentration was < lower limit of quantification).
Measure: Median (Full Range); unit: (μg*day/mL)/respective mg dose
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
(μg*day/mL)/respective mg dose | 2.97 [2.87 to 3.47] | 3.00 [2.43 to 5.36] | 3.48 [2.75 to 4.35]

5. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The median Cmax is presented for each cohort.
Time Frame: Predose (screening), postdose Day 3 to Day 113
Population: as for outcome 4
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
μg/mL | 0.383 [0.317 to 0.387] | 0.764 [0.596 to 1.610] | 2.140 [1.440 to 3.970]

6. Primary Outcome: Median Dose Normalized Cmax
Description: The dose normalized Cmax was calculated for each subject by dividing the parameter by the subject's respective dose in milligrams. The median dose normalized Cmax is presented for each cohort.
Time Frame: Predose (screening), postdose Day 3 to Day 113
Population: as for outcome 4
Measure: Median (Full Range); unit: (μg/mL)/respective mg dose
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
(μg/mL)/respective mg dose | 0.096 [0.079 to 0.097] | 0.076 [0.060 to 0.161] | 0.107 [0.072 to 0.199]

7. Primary Outcome: Median Time to the Maximum Measured Serum Concentration (Tmax)
Description: The median Tmax is presented for each cohort. If the maximum value occurred at more than 1 time point, Tmax was defined as the first time point with this value.
Time Frame: Predose (screening), postdose Day 3 to Day 113
Population: as for outcome 4
Measure: Median (Full Range); unit: day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
day | 14.0 [8.9 to 14.9] | 7.9 [7.0 to 14.9] | 15.0 [6.9 to 16.0]

8. Secondary Outcome: Median Change From Baseline in Visual Acuity for the Study Eye
Description: Best Corrected Visual Acuity (BCVA) letter score was determined using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. The score ranges from 0 to 100 letters, lower number indicating reduced visual acuity; a positive value of change from baseline indicates visual acuity gain and a negative value indicates visual acuity loss.
Time Frame: Day 1 to Day 113
Population: The efficacy set included all subjects who received any amount of the study drug.
Measure: Median (Full Range); unit: letters read correctly
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
letters read correctly | 1 [0 to 4] | 3 [-9 to 11] | -1 [-4 to 10]

9. Secondary Outcome: Median Change From Baseline in Central Retinal Thickness, Central Retinal Lesion Thickness and Central Subfield Thickness in the Study Eye
Description: Central retinal thickness, central retinal lesion thickness and central subfield thickness were determined using Spectral Domain Optical Coherence Tomography (SD-OCT).
Time Frame: Day 1 to Day 113
Population: The safety set included all subjects who received any amount of study drug.
Measure: Median (Full Range); unit: micrometers
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
micrometers
  Retinal thickness | -106 [-129 to 71.5] | 5.0 [-109 to 22.0] | 37.5 [-9.5 to 170.5]
  Retinal lesion thickness | -79.5 [-128 to 64.0] | 2.5 [-104 to 31.5] | 19.0 [-21.5 to 212.0]
  Central Subfield Thickness | -29.0 [-48.0 to 42.0] | -12.0 [-80.0 to 20.0] | 65.0 [-11.0 to 138.0]

10. Secondary Outcome: Median Change From Baseline in Macular Cube Volume in the Study Eye
Description: Macular cube volume was determined using SD-OCT.
Time Frame: Day 1 to Day 113
Population: The safety set included all subjects who received any amount of study drug.
Measure: Median (Full Range); unit: mm^3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 7
mm^3 | -0.4 [-2.1 to 0.2] | -0.1 [-0.3 to 0.2] | 0.3 [-0.3 to 0.7]

ADVERSE EVENTS:
Time Frame: TEAEs were collected from Day 1 up to the final study visit at Day 113 (approximately 16 weeks).
Description: The safety set included all subjects who received any amount of study drug.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=7)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes